CLINICAL TRIAL: NCT02801266
Title: Improving Contraceptive Counseling in the United States
Acronym: ICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Planned Parenthood Federation of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FPRPA006057; 12-9103 (Other: NYU Committee on Activities Involving Human Subjects)
Record Dates: First submitted 2016-06-02; First posted 2016-06-15 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2016-06

CONDITIONS: New Behavioral Protocol; Treatment as Usual
Keywords: Contraception; Reproductive and Sexual Health; Counseling; Contraceptive Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention arm receives contraceptive counseling from counselors who underwent training on the use of evidence informed birth control counseling.
  Interventions: Behavioral: Evidence informed birth control counseling
- No intervention (No Intervention): The no intervention arm receives contraceptive counseling from counselors who underwent no additional training beyond what they normally receive.

INTERVENTIONS:
Behavioral: Evidence informed birth control counseling — Counselors underwent training on the use of 10 best practices for contraceptive counseling.
  Other Names: Improving contraceptive counseling in the United States
  Arms: Intervention

SUMMARY:
This project develops a contraceptive counseling protocol (CCP) grounded in scientific evidence and evaluates the CCP for promoting behaviors conducive to preventing unintended pregnancy among women. The project develops and refines the CCP using focus groups and in-depth interviews with (a) key administrators in the national office of Planned Parenthood (b) key administrators in participating Title X clinics, (c) contraceptive counselors, and (d) clients of the health centers. The CCP uses scientifically grounded principles for guiding effective decision making and provider-client communication. Ten Title X clinics are randomly assigned to one of two conditions (5 clinics per condition): (1) treatment as usual (TAU) or (2) implementation of the CCP. Approximately 150 women are selected for study participation in each clinic, yielding about 1,400 participants (half control and half CCP). Immediately following their counseling session, women complete a computer-administered interview that serves as a fidelity check and permits evaluation of the effects of the CCP on variables associated with counseling satisfaction. All women are re-interviewed by phone 6 months later and 12 months later. The effect of the CCP on method-choice effectiveness, method switching, gaps in protection, and use accuracy are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Must be seeking contraception from clinic on day of recruitment

Exclusion Criteria:

* Not seeking contraception from clinic on day of recruitment

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1418 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with counselors as assessed by 5 point Likert rating scales using questionnaire designed for this study at immediate posttest. | immediately after counseling session
Patient satisfaction with counseling session as assessed by 5 point Likert rating scales using a questionnaire designed for this study at immediate posttest. | immediately after counseling session
Patient satisfaction with clinic experience overall as assessed by 5 point Likert rating scales using a questionnaire designed for this study at immediate posttest. | immediately after counseling session
Patient satisfaction with clinic experience overall as assessed by 5 point Likert rating scales using a questionnaire designed for this study at 6 months. | 6 months from initial clinic visit
Patient satisfaction with clinic experience overall as assessed by 5 point Likert rating scales using a questionnaire designed for this study at 12 months. | one year from initial clinic visit

SECONDARY OUTCOMES:
Type of contraceptive method currently using (including none and dual use) as assessed by a questionnaire designed for this study (e.g., what method of birth control are you currently using). | six months to one year from initial clinic visit

OTHER OUTCOMES:
Method switching for pill users as assessed by a questionnaire designed for this study asking current method used at posttest to determine if it is no longer the pill using questions designed for this study | six months to one year from initial clinic visit
Gaps in pregnancy protection (number of weeks not using any birth control during contraceptive method switches as assessed by a questionnaire designed for this study using retrospective recall | six months to one year from initial clinic visit
Counselor behavior (topics covered during counseling) as assessed by a questionnaire designed for this study asking if counselor did or did not address key topics about method use | six months to one year from initial clinic visit
Pill users retrospective report of the number of missed pills using a questionnaire designed for this study | six months to one year from initial clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: James J Jaccard, PhD, Principal Investigator — New York University
Locations (1):
- New York University, Silver School of Social Work, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No